CLINICAL TRIAL: NCT01031797
Title: QT Dispersion in Patients With Systemic Lupus Erythematosus: the Impact of Disease Activity
Brief Title: QT Dispersion in Patients With Systemic Lupus Erythematosus (SLE)
Status: Completed | Type: Observational
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Javad Kojuri, Shiraz University of medical sciences
Other Study IDs: 86-1256
Record Dates: First submitted 2009-12-12; First posted 2009-12-15 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2007-07

CONDITIONS: SLE
Keywords: SLE; Disease activity score; QT dispersion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- High SLEDAS: High SLE disease activity score
- Low SLEDAS: SLE patient with low score

SUMMARY:
QT dispersion can be a useful, simple noninvasive method for the early detection of cardiac involvement in SLE patients with active disease. The investigators therefore recommend cardiovascular evaluation for every SLE patient with an SLEDAI higher than 10.

DETAILED DESCRIPTION:
Objective: Patients with systemic lupus erythematosus (SLE) have increased cardiovascular morbidity and mortality. Although autopsy studies have documented that the heart is affected in most SLE patients, clinical manifestations occur in less than 10%. QT dispersion is a new parameter that can be used to assess homogeneity of cardiac repolarization and autonomic function. We compared the increase in QT dispersion in SLE patients with high disease activity and mild or moderate disease activity.

Methods: One hundred twenty-four patients with SLE were enrolled in the study. Complete history and physical exam, ECG, echocardiography, exercise test and SLE disease activity index (SLEDAI) were recorded. Twenty patients were excluded on the basis of our exclusion criteria. The patients were divided to two groups based on SLEDAI: 54 in the high-score group (SLEDAI >10) and 50 in the low-score group (SLEDAI <10).

ELIGIBILITY:
Inclusion Criteria:

* no administration of drugs that would potentially influence QT duration except hydroxychloroquine
* no history of ischemic heart disease, congestive heart failure, atrial fibrillation, bundle branch block or abnormal serum electrolytes
* normal resting ECG and a good-quality ECG recording to measure the QT interval.

Exclusion Criteria:

* moderate or severe valve disease
* atrial fibrillation and other ECG abnormalities
* systolic left ventricular dysfunction (ejection fraction <50% or left ventricular end diastolic dimension >5.5 mm
* unreliable identification of the end of the T wave in the ECG and
* known presence of cardiac disease including hypertension, diabetes or coronary artery disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred twenty-four patients with SLE were enrolled in the study. Complete history and physical exam, ECG, echocardiography, exercise test and SLE disease activity index (SLEDAI) were recorded. Twenty patients were excluded on the basis of our exclusion criteria. The patients were divided to two groups based on SLEDAI: 54 in the high-score group (SLEDAI >10) and 50 in the low-score group (SLEDAI <10).
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
QT dispersion

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Kojuri J, Nazarinia MA, Ghahartars M, Mahmoody Y, Rezaian Gr, Liaghat L. QT dispersion in patients with systemic lupus erythematosus: the impact of disease activity. BMC Cardiovasc Disord. 2012 Feb 27;12:11. doi: 10.1186/1471-2261-12-11. PMID 22369270